CLINICAL TRIAL: NCT01708785
Title: Learning Theory to Improve Obesity Treatment (Intervention for Regulation of Cues)
Brief Title: Learning Theory to Improve Obesity Treatment
Acronym: iROC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kerri Boutelle, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 120431; 1R01DK094475-01A1 (NIH)
Record Dates: First submitted 2012-10-11; First posted 2012-10-17 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: obesity; overweight; overweight children; overweight parents; overeating; eating in the absence of hunger; families with overweight child; body mass index; BMI; weight; childhood obesity; treatment; cue exposure treatment; cravings; habituation to food cues; psychophysiological response to food cues; intervention; experiments; family based treatment; behavioral treatment
MeSH Terms: conditions — Obesity; Overweight; Hyperphagia; Body Weight; Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Single context (Active Comparator): Subjects will be exposed to food cues in a single context.
  Interventions: Behavioral: Partial Reinforcement - Enhanced Cue Exposure Treatment; Behavioral: Partial Reinforcement -Consistent Cue Exposure Treatment
- Multiple contexts (Experimental): Subjects will be exposed to food cues in multiple contexts.
  Interventions: Behavioral: Partial Reinforcement - Enhanced Cue Exposure Treatment; Behavioral: Partial Reinforcement -Consistent Cue Exposure Treatment
- 8 treatment sessions (Active Comparator): Subjects receive 8 treatment sessions.
  Interventions: Behavioral: Single food Cue Exposure Treatment; Behavioral: Multiple food Cue Exposure Treatment
- 16 treatment sessions (Experimental): Subjects receive 16 treatment sessions
  Interventions: Behavioral: Single food Cue Exposure Treatment; Behavioral: Multiple food Cue Exposure Treatment

INTERVENTIONS:
Behavioral: Single food Cue Exposure Treatment — Subjects will be exposed to the same set of 4 foods in each cue exposure treatment session.
  Arms: 16 treatment sessions; 8 treatment sessions
Behavioral: Multiple food Cue Exposure Treatment — Subjects will be exposed to a different set of 4 foods in each cue exposure treatment session.
  Arms: 16 treatment sessions; 8 treatment sessions
Behavioral: Partial Reinforcement - Enhanced Cue Exposure Treatment — Subjects will take random additional tastes of the food during cue exposure treatment.
  Arms: Multiple contexts; Single context
Behavioral: Partial Reinforcement -Consistent Cue Exposure Treatment — Subjects will consistently take the same tastes of the food during cue exposure treatment.
  Arms: Multiple contexts; Single context

SUMMARY:
The purpose of this study is to optimize an obesity treatment program targeting overweight 8-12 year old children using "Cue Exposure Training".

DETAILED DESCRIPTION:
The goal of the Cue Exposure program is to train children to resist cues to eat unhealthy foods. Through a series of experimental studies, the investigators will evaluate how many weekly treatment visits there should be, whether children should be exposed to a single food or multiple foods during treatment, whether to use partial reinforcement or not, whether visits should be daily or weekly, and whether the exposures should be in single or multiple contexts. The investigators will be recruiting parent-child dyads in the San Diego community to participate in 8 to 16 weekly or daily treatment sessions either in their home, community center, or our lab, depending on the treatment arm. Parents and children will complete baseline and post-treatment assessments consisting of collecting psychophysiological data, completing laboratory tasks, and completing questionnaires. The investigators will be evaluating which treatment condition reduces overeating (as measured by our laboratory tasks).

ELIGIBILITY:
Inclusion Criteria:

* Response to an advertisement for the study,
* An overweight or obese child in the family who is between the ages of 8 and 13,
* The 8-13 year old child must be above the 85th BMI % for age and gender,
* Parent willing to participate and attend all meetings,
* Parent who can read at a minimum of a 5th grade level in English,
* Parent and child willing to commit to attendance and assessments,
* Child who eats in the absence of hunger.

Exclusion Criteria:

* Major child psychiatric disorder diagnoses,
* An obese child over the 99.9th BMI %
* Child or parent diagnoses of diabetes for which physician supervision of diet is needed or diagnosis of serious current physical diseases (such as cancer, multiple sclerosis, lupus) which could significantly decrease their ability to participate in the intervention (parent report),
* Child taking a medication that can affect cognitive functioning, such as attention, concentration, or mental status.
* Family with restrictions on types of food, such as food allergies, or religious or ethnic practices that limit the foods available in the home (these restrictions affect their ability participate in the food exposures because it would limit the variety of foods available to do exposures with),
* Child with an active eating disorder (based on parent and child self-report)
* Major parent psychiatric or eating disorder.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2012-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in overeating (Eating in the absence of hunger) from baseline at an average of 3 months and 6 months | Change from baseline at an average of 3 months and 6 months
  Reduce overeating or eating in the absence of hunger in response to food cues. Habituation to food cues.
Change in child weight | Change from baseline at an average of 3 and 6 months
  BMI, BMIz

SECONDARY OUTCOMES:
Change in parent weight from baseline at average of 3 and 6 months | Change from baseline at average of 3 and 6 months
  Measured by BMI (Body Mass Index)
Change in attention to food cues from baseline at average of 3 and 6 months | Change from baseline at average of 3 and 6 months
  Reduce attention to food cues, redirect attention to neutral (non-food cues). Measured by computer program measuring response time
Change in impulsivity/Inhibition from baseline at average of 3 and 6 months | Change from baseline at average of 3 and 6 months
  Reduce impulsive behavior response to both food and non-food cues. Measured by behavioral tasks
Change in psychophysiological measures of responsivity to food cues from baseline at average of 3 and 6 months | Change from baseline at average of 3 and 6 months
  Salivation/swallowing using EMG (electromyography), skin conductance, heart rate and heart rate variability.
Change in level of self-reported cravings in response to palatable food cues from baseline at average of 3 and 6 months | Change from baseline at average of 3 and 6 months
  Participants will rate their cravings on a scale of 1-10.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, Ph.D., Principal Investigator — UCSD
Locations (1):
- Center for Health Eating and Activity Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boutelle KN, Zucker NL, Peterson CB, Rydell SA, Cafri G, Harnack L. Two novel treatments to reduce overeating in overweight children: a randomized controlled trial. J Consult Clin Psychol. 2011 Dec;79(6):759-71. doi: 10.1037/a0025713. PMID 22122291
- [Background] Epstein LH, Myers MD, Raynor HA, Saelens BE. Treatment of pediatric obesity. Pediatrics. 1998 Mar;101(3 Pt 2):554-70. PMID 12224662
- [Background] Nederkoorn C, Smulders FT, Jansen A. Cephalic phase responses, craving and food intake in normal subjects. Appetite. 2000 Aug;35(1):45-55. doi: 10.1006/appe.2000.0328. PMID 10896760
- [Background] Nederkoorn C, Jansen A. Cue reactivity and regulation of food intake. Eat Behav. 2002 Spring;3(1):61-72. doi: 10.1016/s1471-0153(01)00045-9. PMID 15001020